

# TRIAL STATISTICAL ANALYSIS PLAN MODULE C (BI 754091+ BI 836880)

c39700100-01

**BI Trial No.:** 1381.9

**Title:** An open-label, Phase II trial evaluating the safety and efficacy of

BI 836880 in combination with ezabenlimab in PD-(L)1 na\"ive and

PD-(L)1 pretreated patient populations with advanced and/or

metastatic solid tumours who have had at least one line of systemic

therapy

Investigational

Ezabenlimab (BI 754091 [anti-PD-1])

**Product(s):** 

BI 836880 (anti-VEGF/Ang2)

Responsible trial statistician(s):

Phone:

Date of statistical analysis plan:

20 JUL 2022 SIGNED

**Version:** Final


#### Proprietary confidential information

© 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

**7.8.2** 

7.8.3

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1. | TABLE OF CONTENTS |
|----------------|--------------------------------------------------|
| TITLE PA | AGE1 |
| 1. | TABLE OF CONTENTS2 |
| LIST OF | ΓABLES |
| 2. | LIST OF ABBREVIATIONS5 |
| 3. | INTRODUCTION6 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY7 |
| 5. | ENDPOINT(S)8 |
| 5.1 | PRIMARY ENDPOINT(S)8 |
| <b>5.2</b> | SECONDARY ENDPOINT(S) |
| 5.2.1 | Key secondary endpoint(s)8 |
| 5.2.2 | Secondary endpoint(s)8 |
| 5.4.1 | Demographics and baseline characteristics8 |
| <b>6.</b> | GENERAL ANALYSIS DEFINITIONS |
| 6.1 | TREATMENT(S) |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS |
| 6.3 | SUBJECT SETS ANALYSED11 |
| 6.5 | POOLING OF CENTRES11 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS11 |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS11 |
| 7. | PLANNED ANALYSIS14 |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS14 |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION14 |
| 7.3 | TREATMENT COMPLIANCE |
| 7.4 | PRIMARY ENDPOINT(S) |
| 7.4.1 | Primary analysis |
| 7.4.2 | Interim analysis 14 |
| 7.5<br>7.5.1 | SECONDARY ENDPOINT(S) |
| 7.5.1<br>7.5.2 | (Other) Secondary endpoint(s) |
| 1.0.4 | (Other) becomes y emponings, |
| 7.7 | EXTENT OF EXPOSURE |
| <b>7.8</b> | SAFETY ANALYSIS |
| 7.8.1 | Adverse events15 |

## LIST OF TABLES

| Table 6.2: 1 | Module C Important protocol deviations | 10 |
|---|---|---|
| Table 6.7: 1 | Nominal time points and windows for imaging | 12 |
| Table 6.7: 2 | Time windows for assignment of safety lab measurements to visits for statistical analysis | 12 |
| Table 6.7: 3 | Time windows for patients discontinuing treatment before Cycle 16 or receive treatment beyond Cycle 16 | |
| Table 10: 1 | History table | 22 |

#### 2. LIST OF ABBREVIATIONS

| Term | Definition / description |
|--------|-----------------------------------------------|
| AE | Adverse Event |
| BHM | Bayesian Hierarchical Model |
| CR | Complete Response |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| DC | Disease Control |
| DoR | Duration of Response |
| ICH | International Conference on Harmonisation |
| IPD | Important Protocol Divations |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MQRM | Medical Quality Review Meeting |
| MTD | Maximum Tolerated Dose |
| OR | Objective Response |
| OS | Overall Survival |
| PD | Progression of Disease |
| PFS | Progression-Free Survival |
| PK | Pharmacokinetics |
| PR | Partial Response |
| PSTAT | Project Statistician |
| PT | Preferred Term |
| RECIST | Response Evaluation Criteria in Solid Tumours |
| REP | Residual Effect Period |
| SA | Statistical Analysis |
| SAE | Serious Adverse Event |
| SD | Stable Disease |
| SOC | System Organ Class |
| ToC | Table of Contents |
| TS | Treated Set |
| TSAP | Trial Statistical Analysis Plan |

**** 

Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3. INTRODUCTION

As per ICH E9 [1], the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the Master and Module C Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the Module C TSAP is based on the planned analysis specification as written in Master and Module C CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, Module C TSAP readers may consult the Master and Module C CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomization.

SAS® Version 9.4 or the latest version will be used for analyses.

R v3.5.1 and JAGS v4.3.0 or the latest versions will be used for BHM analysis.

#### CHANGES IN THE PLANNED ANALYSIS OF THE STUDY 4.

Refer to the Master TSAP.

## 5. ENDPOINT(S)

## **5.1 PRIMARY ENDPOINT(S)**

Refer to the Master TSAP.

## 5.2 SECONDARY ENDPOINT(S)

## 5.2.1 Key secondary endpoint(s)

This section is not applicable because no key secondary endpoints have been defined in the CTP.

## 5.2.2 Secondary endpoint(s)

Refer to the Master TSAP.

## **5.3 FURTHER ENDPOINT(S)**

Refer to the Master TSAP.

## 5.4.1 Demographics and baseline characteristics

Refer to the Master TSAP.





#### 6. GENERAL ANALYSIS DEFINITIONS

## 6.1 TREATMENT(S)

Patients in this Module of the clinical trial will receive BI 836880 combined with BI 754091 by i.v. infusion after signing the Master and Module C informed consent forms and completing the screening processes. Treatment will be administered every 3 weeks (1 cycle = 21 days).

For definition of treatment periods refer to the Master TSAP.

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Refer to master TSAP for definition of iPD criteria listed in Table 6.2: 1. The module C specific iPD criteria are listed in <u>Table 6.2: 1</u> below.

Table 6.2: 1 Module C Important protocol deviations

| Category /<br>Code | | Description | Comment /<br>Example | Excluded from | Automatic/<br>Manual |
|---|---|---|---|---|---|
| A | | Entrance criteria not met | | | |
| | Ala | Inclusion criteria not met | | | |
| | Ala.1 | No measurable lesions according to RECIST 1.1 | Inclusion criterion (IN) 3 not met | None | Automatic |
| | A2a | <b>Exclusion criteria met</b> | | | |
| | A2a.1 | Unresolved toxicity from previous treatment. | Exclusion criterion (EX) 2 met | None | Automatic |
| | A2a.2 | Significant cardiovascular/ cerebrovascular disease. | Exclusion criterion (EX) 3 met | None | Automatic |
| | A2a.3 | Severe haemorrhagic or<br>thromboembolic event<br>in past 12 months | Exclusion criterion (EX) 4 met | None | Automatic |
| | A2a.4 | Known inherited predisposition to bleeding or to thrombosis | Exclusion criterion (EX) 5 met | None | Automatic |
| | A2a.5 | Patients who require full-dose anticoagulation | Exclusion criterion (EX) 6 met | None | Automatic |
| | A2a.6 | Prior anti-angiogenic<br>therapy (with the<br>exception of CRC<br>Cohort) | Exclusion criterion (EX) 7 met | None | Automatic |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6.3 SUBJECT SETS ANALYSED

#### Module C Screened Set:

This patient set includes all patients who have signed the informed consent for the study and module C. The screened set will be used for patient disposition tables.

#### Module C Treated Set (TS):

This patient set includes all patients who were documented to have received at least one dose of trial medications in Module C. The TS is used for both efficacy analysis and safety analyses.

## Module C Pharmacokinetic Set (PKS):

This patient set includes all patients in the TS with at least one valid plasma concentration. PKS will be used for all pharmacokinetic analyses.



#### 6.5 POOLING OF CENTRES

This section is not applicable because centre/country is not included in the statistical analyses.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Refer to the Master TSAP.

#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Baseline values will be the measurements taken most recently prior to first administration of study drug in Module C.

Study day will be calculated relative to the date of the first administration of study drug in Module C. The day prior to first administration of study drug will be 'Day -1' and the day of first administration of study drug will be 'Day 1'; therefore 'Day 0' will not exist.

In order to identify whether consecutive imaging time points are missing for a given patient in this module, a nominal time point (i.e. Week 6, 12, 18 ... etc.) will be assigned to each and every image. This is achieved by creating windows for every radiological response assessment. These windows are defined in <u>Table 6.7: 1</u>.

Table 6.7: 1 Nominal time points and windows for imaging

| Nominal time point (weeks from start of study drug) | Due date of scans (days)* | Window (days) |
|---|---|---|
| 6 | 43 | 1 to ≤ 64 |
| 12 | 85 | 65 to ≤ 106 |
| 18 | 127 | $107 \text{ to} \le 148$ |
| 24 | 169 | 149 to $\leq$ 200 |
| 33 | 232 | 201 to ≤ 263 |
| 42 | 295 | 264 to ≤ 326 |
| 51 | 358 | 327 to ≤ 389 |
| Etc., 9-week interval | Etc. | Etc. |

<sup>\*</sup> The date of the first dose of study medication is Day 1

If a patient does not have an image in one of the windows described above, he/she will be said to have missed an assessment for that time point.

Table 6.7: 2 Time windows for assignment of safety lab measurements to visits for statistical analysis

| Window No. | Nominal visit | Nominal day | Interval |
|---|---|---|---|
| 0 | Cycle 1 | 1 | NA |
| 1 | Cycle 1 | 8 | [2,11] |
| 2 | Cycle 1 | 15 | [12,18] |
| 3 | Cycle 2 | 22 | [19,32] |
| 4 | Cycle 3 | 43 | [33,53] |
| n+1 | Cycle n | 21*(n-1)+1 | [21*(n-1)-9,<br>21*(n-1)+11] |
| 18 | EOT | 21*16+1 | [327, 351] |
| 19 | Safety Follow<br>up | 21*16+31 | [352, ∞] |

Note: n=3,4,5,...,16.


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For patients discontinuing treatment before Cycle 16 or receive treatment beyond Cycle 16, identify the last treatment cycle n (>=3) and time windows of EOT and Safety Follow up will be derived according to Table 6.7: 3.

Table 6.7: 3 Time windows for patients discontinuing treatment before Cycle 16 or receive treatment beyond Cycle 16

| Window No. | Nominal visit | Nominal day | Interval |
|---|---|---|---|
| n+1 | Cycle n | 21*(n-1)+1 | [21*(n-1)-9,<br>21*(n-1)+11] |
| n+2 | ЕОТ | 21*n+1 | [21*n-9,<br>21*n+15] |
| n+3 | Safety Follow<br>up | 21*n+31 | [21*n+16, ∞] |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7. PLANNED ANALYSIS

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Refer to the Master TSAP.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Refer to the Master TSAP.

#### 7.3 TREATMENT COMPLIANCE

Only descriptive statistics are planned for this section.

### 7.4 PRIMARY ENDPOINT(S)

## 7.4.1 Primary analysis

Refer to the Master TSAP for BHM [2] approach description for the primary analysis of ORR.

For the BHM approach, a non-informative normal distribution with mean 0 and standard deviation of 2 is specified for the mean  $\mu$ . For the inter-cohort heterogeneity parameter  $\tau$ , a half normal distribution with parameter 1 is used which is a very conservative assumption regarding between-cohort variability and hence leads to only little borrowing of data across patient cohorts because there is little prior information on the strength of the correlation between the treatment effects across cohorts in Module C.

Prior to the primary analysis, the interim futility analysis is planned (section 7.4.2).

## 7.4.2 Interim analysis

Interim analysis will be performed when deemed necessary. Final/primary analysis for a specific treatment combination or cohort will be considered as interim analysis. A cohort or Module may be closed, if determined to be appropriate based on results of interim analyses. Note that interim analysis will not lead to any modifications within the running trial unless otherwise stated in a Module.

Refer to section 7.4 of the Master protocol and Module C protocol for details.

## 7.5 SECONDARY ENDPOINT(S)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.5.1 Key secondary endpoint(s)

This section is not applicable because no key secondary endpoints have been defined in the CTP.

## 7.5.2 (Other) Secondary endpoint(s)

Refer to the Master TSAP.



#### 7.7 EXTENT OF EXPOSURE

The numbers of cycle initiated will be summarized descriptively for each cohort.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the treated set (TS). Analysis will be performed as defined in Section 7.3.4 of the CTP.

## 7.8.1 Adverse events

Refer to the Master TSAP.

## 7.8.2 Laboratory data

Refer to the Master TSAP.

## 7.8.3 Vital signs

Refer to the Master TSAP.

### 7.8.4 ECG

N/A

#### **7.8.5** Others

## 7.8.5.1 PK parameters

For ezabenlimab as well as for BI 836880 actual sampling times will be listed. Raw concentration values will be summarized descriptively per nominal time point. The derived PK parameters will be summarized descriptively.

As described in Section 5.3.1 of the Module C CTP, plasma concentration values will be used to support an exploratory model based analysis, using pooled data from other studies. These analyses will be done and reported outside of the CTR.





## 8. REFERENCES

- 1. CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version.
- 2. Berry SM, Broglio KR, Groshen S, Berry DA. Bayesian hierarchical modeling of patient subpopulations: Efficient designs of Phase II oncology clinical trial. Clinical Trials 10 (5), 720-734 (2013) [R18-2260].



#### **HISTORY TABLE 10.**

History table Table 10: 1

| - | Version | Date<br>(DD-MMM-<br>YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|---|
| | Final | DD-MMM-YY | | None | This is the final TSAP |



#### APPROVAL / SIGNATURE PAGE

Document Number: c39700100 Technical Version Number: 1.0

**Document Name:** 08-01-tsap-module-c-core1

**Title:** An open-label, Phase II trial evaluating the safety and efficacy of BI 836880 in combination with ezabenlimab in PD-(L)1 naïve and PD-(L)1 pretreated patient populations with advanced and/or metastatic solid tumours who have had at least one line of systemic therapy

## Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|--------------------------------|-----------|------------------------|
| Author | | 04 Aug 2022 15:43 CEST |
| Approval-Biostatistics | | 04 Aug 2022 15:47 CEST |
| Approval-Team Member Medicine | | 04 Aug 2022 15:52 CEST |
| Approval-Clinical Trial Leader | | 12 Aug 2022 17:30 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c39700100Technical Version Number:1.0

## (Continued) Signatures (obtained electronically)

| Meaning of Signature Signed by Date Signed |
|--------------------------------------------|
|--------------------------------------------|